CLINICAL TRIAL: NCT06936761
Title: Comparison of Two Induction Methods in Awake Extubated Children at Risk for Respiratory Adverse Events: A Retrospective Study
Brief Title: This Study Evaluated the Safety of Awake Extubation in Children at Risk for Respiratory Events Undergoing General Anesthesia.
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, FUNDA ARUN, Assis. Prof., Selcuk University
Other Study IDs: F005; 07/2024 (Other: Selcuk University ethical commitee)
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Tract Infection
Keywords: awake extubation; general anesthesia; children; sevoflurane
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Sevoflurane (8% in oxygen 2% and air 2%): Inhaler induction with sevoflurane 8% in oxygen 2% and air 2%, intravenous induction with propofol (3-5 mg/kg)
  Interventions: Drug: Sevoflurane
- propofol (3-5 mg/kg IV): This is a retrospective study about rottenly used anesthesia drugs.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — This is an observational study about routines of anesthesia induction and extubation
  Groups: propofol (3-5 mg/kg IV)
Drug: Sevoflurane — This is a retrospective evolution of anesthesia drugs used routinely in an anesthesia clinic.
  Other Names: propofol
  Groups: Sevoflurane (8% in oxygen 2% and air 2%)

SUMMARY:
The primary aim of this study was to evaluate the safety of awake extubation in children at risk for PRAEs undergoing general anesthesia. Specifically, this study seeks to compare the effects of sevoflurane and propofol induction on postoperative (emergence and recovery) respiratory outcomes in these patients. This study aims to provide insights that could enhance anesthesia protocols in pediatric populations with heightened respiratory risks by identifying potential differences in airway-related adverse events between the two agents.

DETAILED DESCRIPTION:
Awake extubation is advantageous in ambulatory settings where patients are discharged on the same day, as it reduces the risk of airway-related complications during recovery and ensures a smoother transition to postoperative care. When children come in for dental treatments requiring GA, they can face higher chances of respiratory issues due to things like colds, asthma, or unique physical traits. The way we introduce anesthesia is important in helping prevent these complications. In this context, sevoflurane and propofol are two commonly used agents for the induction of anesthesia in children. Sevoflurane, a volatile anesthetic agent, is favored for its non-irritating nature and smooth induction process, particularly in pediatric patients. However, its use has been associated with a higher incidence of airway complications, including laryngospasm and coughing. On the other hand, propofol, a widely used intravenous (IV) agent, is known for its rapid onset and favorable recovery profile. It also reduces airway reflex responses, potentially decreasing the risk of respiratory complications during induction and emergence.

Current evidence suggests that extubating during emergence from anesthesia does not significantly alter clinical outcomes for healthy children. A large prospective cohort study examined a population at particularly high risk for perioperative respiratory adverse events (PRAEs). Additionally, a detailed analysis of the risk factors within the cohort suggested that the timing of extubation seemed to impact the occurrence of laryngospasm and severe complications of coughing.

The primary aim of this study was to evaluate the safety of awake extubation in children at risk for PRAEs undergoing general anesthesia. Specifically, this study seeks to compare the effects of sevoflurane and propofol induction on postoperative (emergence and recovery) respiratory outcomes in these patients. By identifying potential differences in airway-related adverse events between the two agents, this study aims to provide insights that could enhance anesthesia protocols in pediatric populations with heightened respiratory risks.

All children were extubated while awake when they demonstrated facial grimacing, adequate tidal volumes, an appropriate respiratory rate, coughing with an open mouth, opening their eyes, and purposeful movements. The anesthesiologist placed all children on 100% oxygen prior to extubation and transported them in the lateral position to the Post-Anesthesia Care Unit (PACU) after ensuring they could maintain adequate airway patency. Oxygen saturation was continuously monitored until discharge from the PACU. Room air was administered unless saturation fell below 95%, at which point supplemental oxygen was provided. All incidents of laryngospasm, bronchospasm (serious risk factors; I, II), desaturation below 95%, airway obstruction, severe coughing, or postoperative stridor (minor risk factors; III, IV) were recorded, along with any airway interventions. The primary outcome measure for analysis was oxygen saturation below 95% for more than 10 seconds. However, shorter desaturation episodes were also captured since oxygen saturation was continuously recorded per institutional guidelines. Any treatment required in response to respiratory adverse events was documented.

Subsequently, the responsible anesthesiologist gathered and reviewed all relevant data from anesthesia and PACU records. Patients with known cardiac disease, airway, or thoracic malformations were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* At least have one criteria of the ISAAC questionnaire
* ASA1&2

Exclusion Criteria:

* cardiac disease
* airway or thoracic malformations
* ASA3

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 425 children (aged 2 to 13) underwent elective dental rehabilitation under general anesthesia.
  During preoperative anesthesia evaluations, an anesthesia research nurse who was unaware of the study protocol administered a modified ISAAC (International Study of Asthma and Allergies in Childhood) questionnaire. The presence of one or more risk factors for PRAEs was recorded, including a cold or flu within the previous two weeks, wheezing more than three times in the past 12 months, wheezing during exercise, dry nocturnal cough, current or past eczema, two family members with asthma, two family members with eczema, two family members with hay fever, and smoking by the mother or both parents.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome was defined as a drop in oxygen saturation (SpO₂) below 95% lasting longer than 10 seconds. | 10 sec
  Room air was administered unless saturation fell below 95%, at which point supplemental oxygen was provided.
Serious risk factors (in ASA I and II patients): Laryngospasm Bronchospasm | 3 Hours in PACU
Minor Risk factors: Airway obstruction Severe coughing Postoperative stridor | 3 Hours in PACU

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Faculty of Dentistry, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No